CLINICAL TRIAL: NCT00162786
Title: Comparative Effects of Rupatadine 10 mg, Hydroxyzine 50 mg and Placebo on Actual Driving Performance
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DM02RUP/IV/04
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2005-12

CONDITIONS: Healthy
Keywords: Driving performance; Antihistamine
MeSH Terms: interventions — rupatadine; Hydroxyzine

INTERVENTIONS:
Drug: Rupatadine
Drug: Hydroxyzine
Drug: Placebo

SUMMARY:
The primary objective of this study is to measure and compare the acute effects of rupatadine 10 mg, relative to placebo and hydroxyzine 50 mg as an active control on healthy volunteers' performance on a standard over-the-road driving test and a car-following test.

DETAILED DESCRIPTION:
The study shall be conducted according to a three-way, double-blind, placebo and active controlled crossover design. Treatment groups are identified as follows.

* Rupatadine
* Hydroxyzine
* Placebo

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy males or females
2. Subjects must be experienced drivers.
3. Vision: normal binocular acuity, corrected, or uncorrected.

Exclusion Criteria:

1. Pregnant or nursing females.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-05; Study Completion 2005-11

PRIMARY OUTCOMES:
Actual driving performance

SECONDARY OUTCOMES:
Daytime sleepiness
Subjective sleepiness
Alertness

CONTACTS AND LOCATIONS:
Overall Officials: Erik Vuurman, PhD, Principal Investigator — Maastricht University, Brain and Behaviour Institute
Locations (1):
- Brain and Behaviour Institute, Maastricht, Netherlands